CLINICAL TRIAL: NCT06958536
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo Controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of SAR442970 in Adults With Moderate to Severe Crohn's Disease
Brief Title: A Study to Investigate Efficacy and Safety of SAR442970 in Patients With Crohn's Disease
Acronym: CHROMA CD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRI18450; U1111-1306-7510 (Other: WHO); 2024-517016-30-00 (EU CTIS Number); DRI18450 (Other: Sanofi)
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR442970 Dose Regimen A (Experimental): Participants will receive SAR442970 dose regimen A
  Interventions: Drug: SAR442970
- SAR442970 Dose Regimen B (Experimental): Participants will receive SAR442970 dose regimen B
  Interventions: Drug: SAR442970
- Placebo (Placebo Comparator): Participants will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR442970 — Route of Administration: Subcutaneous
  Arms: SAR442970 Dose Regimen A; SAR442970 Dose Regimen B
Drug: Placebo — Route of Administration: Subcutaneous
  Arms: Placebo

SUMMARY:
This is a phase 2b, randomized, double-blind, 3-arm study for the treatment of Crohn's disease. The primary objective of this study is to assess the efficacy of different doses of SAR442970 compared with placebo in participants with moderate to severe Crohn's disease. The total study duration is up to 168 weeks, with a treatment period of up to 158 weeks including an open-label (OL) long-term extension (LTE) period of up to 104 weeks for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's Disease (CD) for at least 3 months prior to screening
* Confirmed diagnosis of moderate-to-severe CD
* History of prior exposure to standard treatment (5-Amino Salicylates (5-ASAs), steroids, immunomodulators or antibiotics) or advanced therapies (ATs) (biologics or small molecules), but having inadequate response to, loss or response to or intolerance to at least one of these therapies
* On stable doses of standard treatments prior to screening (Oral 5-ASA compounds, Oral corticosteroids, Azathioprine (AZA), 6-Mercaptopurine (6-MP), or Methotrexate (MTX), or Antibiotics, etc.)
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Participants with active Ulcerative Colitis (UC), indeterminate colitis, adenomatous colonic polyps not excised, colonic mucosal dysplasia (low- or high-grade dysplasia) or short bowel syndrome
* Participants with CD isolated to the stomach, duodenum, jejunum, or perianal region, without colonic or ileal involvement
* Participants with following ongoing known complications of CD:

  * Any manifestation that might require bowel surgery while enrolled in the study
  * Participant with ostomy or ileoanal pouch
  * Participant diagnosed with conditions that could interfere with drug absorption including but not limited to short bowel syndrome
  * Participant with surgical bowel resection within the past three months prior to screening, or a history of >3 bowel resections
* History of any other condition which, in the opinion of the Investigator, would put the participant at risk by participation in the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2029-10-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieve endoscopic response at Week 16 | From Baseline to Week 16
  Endoscopic response is defined as decrease in Simple Endoscopic Score for Crohn's Disease (SES-CD) >50% from baseline (or a decrease of at least 2 points for subjects with a baseline score of 4 or more and isolated ileal disease) based on central reading. The SES-CD evaluates 4 endoscopic variables (ulcer size, ulcerated surface, affected surface, and narrowing, each on a scale from 0 (none) to 3 in 5 segments assessed during ileocolonoscopy. The total score is the sum of the 4 endoscopic variable scores and ranges from 0 to 56, where higher scores indicate more severe disease.

SECONDARY OUTCOMES:
Percentage of participants who achieve clinical remission based on Crohn's Disease Activity Index (CDAI) at Week 16 | At Week 16
  CDAI clinical remission is defined as CDAI score <150. CDAI is a composite instrument that includes participant symptoms evaluated over 7 days (abdominal pain, stool frequency and general well-being), as well as presence of complications (arthritis/arthralgia, iritis/uveitis, erythema nodosum/pyoderma gangrenosum/aphthous stomatitis, anal fissure/fistula/abscess, other fistula, and fever), the use of antidiarrheal medicines, presence of an abdominal mass, hematocrit, and body weight. These items are scored individually, weighted, and do not contribute equally to the overall score. The CDAI is derived from summing up the weighted individual scores of eight items. CDAI approximately ranges from 0 to 600 with higher scores indicating more severe disease.
Percentage of participants who achieve PRO-2 (Patient Reported Outcome) clinical remission at Week 16 | At Week 16
  PRO-2 clinical remission is defined as using the average daily Stool Frequency (SF) ≤3 and not worse than baseline and average daily AP ≤1 and not worse than baseline.
Percentage of participants who achieve endoscopic remission based on centrally read SES-CD at Week 16 | At Week 16
  Endoscopic remission is defined as SES-CD ≤4 and at least 2 point reduction versus baseline and no subscore >1 in any individual variable based on central reading.
Percentage of participants who achieve both clinical remission based on CDAI score and endoscopic response based on SES- CD at Week 16 | At Week 16
  CDAI clinical remission is defined as CDAI score <150, endoscopic response is defined as a decrease in SES-CD >50% from baseline (or a decrease of at least 2 points for subjects with a baseline score of 4 or more and isolated ileal disease) based on central reading.
Percentage of participants who achieve CDAI clinical response at Week 16 | At Week 16
  CDAI clinical response is defined as reduction of CDAI ≥100 points from baseline.
Change from baseline in the Inflammatory Bowel Disease Questionnaire (IBDQ) score | From Baseline to Week 16
  The Inflammatory Bowel Disease Questionnaire (IBDQ) is a 32-item instrument assessing health-related quality of life in IBD patients across four dimensions: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). Each question evaluates experiences over the previous two weeks on a 7-point Likert scale from 1 (worst) to 7 (best). The total score ranges from 32 to 224, with higher scores indicating better quality of life. Both domain-specific and overall scores can be calculated.
Change from baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) score | From Baseline to Week 16
  The FACIT-F questionnaire assesses fatigue associated with anemia through 13 fatigue-related questions. Each item is scored on a 5-point Likert scale (0="not at all" to 4="very much"), with total scores ranging from 0 to 52. High scores represent less fatigue. For Crohn's Disease patients, a 7-10 point improvement on the FACIT-F total score may represent meaningful improvements.
On-treatment serum concentrations of SAR442970 at predefined timepoints | Up to End of Study (approximately 164 weeks)
Number and percentage of participants with any Treatment Emergent Adverse Events (TEAEs) during induction, maintenance and Long-term Extension (LTE) treatment period | Up to End of Study (approximately 164 weeks)
Number and percentage of participants with any TEAEs during open-label treatment period | Up to Week 52
Incidence of Anti-drug Antibodies (ADAs) over time | Up to End of Study (approximately 164 weeks)
Percentage of participants who achieve endoscopic remission based on centrally read SES-CD at Week 52 | At Week 52
  Endoscopic remission is defined as SES-CD ≤4 and at least 2 point reduction versus baseline and no subscore >1 in any individual variable based on central reading.
Percentage of participants achieving CDAI clinical remission at Week 52 | At Week 52
  CDAI clinical remission is defined as CDAI <150.
Percentage of participants achieving CDAI clinical remission at both Week 16 and at Week 52 | At Week 52
  CDAI clinical remission is defined as CDAI <150.
Percentage of participants who achieve endoscopic response at Week 52 | At Week 52
  Endoscopic response is defined as decrease in SES-CD >50% from baseline (or a decrease of at least 2 points for subjects with a baseline score of 4 or more and isolated ileal disease) based on central reading.
Percentage of participants who achieve endoscopic response at both Week 16 and Week 52 | At Week 52
  Endoscopic response is defined as decrease in SES-CD >50% from baseline (or a decrease of at least 2 points for subjects with a baseline score of 4 or more and isolated ileal disease) based on central reading.
Percentage of participants who achieve CDAI clinical response at Week 52 | At Week 52
  CDAI clinical response is defined as reduction of CDAI ≥100 points from baseline.
Percentage of participants who achieve both clinical remission based on CDAI score and endoscopic response based on SES- CD at Week 52 | At Week 52
  CDAI clinical remission is defined as CDAI score <150, endoscopic response is defined as a decrease in SES-CD >50% from baseline (or a decrease of at least 2 points for subjects with a baseline score of 4 or more and isolated ileal disease) based on central reading.

CONTACTS AND LOCATIONS:
Locations (56):
- United States (16):
  - Investigational Site Number: 8400005, Escondido, California
  - Investigational Site Number: 8400001, Lancaster, California
  - Investigational Site Number: 8400017, Kissimmee, Florida
  - Investigational Site Number: 8400015, Lighthouse PT, Florida
  - Investigational Site Number: 8400012, Miami, Florida
  - Investigational Site Number: 8400011, Palmetto Bay, Florida
  - Investigational Site Number: 8400019, Marietta, Georgia
  - Investigational Site Number: 8400025, Iowa City, Iowa
  - Investigational Site Number: 8400022, Boston, Massachusetts
  - Investigational Site Number: 8400008, Wyoming, Michigan
  - Investigational Site Number: 8400013, St Louis, Missouri
  - Investigational Site Number: 8400002, Chapel Hill, North Carolina
  - Investigational Site Number: 8400009, Harrisburg, Pennsylvania
  - Investigational Site Number: 8400002, Fredericksburg, Texas
  - Investigational Site Number: 8400016, Ogden, Utah
  - Investigational Site Number: 8400027, Richmond, Virginia
- Australia (3):
  - Investigational Site Number: 0360002, Brisbane, Queensland
  - Investigational Site Number: 0360004, Kurralta Park, South Australia
  - Investigational Site Number: 0360001, Footscray
- Investigational Site Number: 0560001, Leuven, Belgium
- China (6):
  - Investigative Site: 1560003, Changsha
  - Investigative Site: 1560005, Changzhou
  - Investigational Site Number: 1560001, Guangzhou
  - Investigational Site Number: 1560006, Hangzhou
  - Investigative Site: 1560004, Nanchang
  - Investigative Site: 1560002, Shanghai
- Czechia (2):
  - Investigational Site Number: 2030002, Brno, JM
  - Investigational Site Number: 2030003, Hradec Králové
- France (3):
  - Investigational Site Number: 2500001, Montpellier
  - Investigative Site: 2500003, Nice
  - Investigational Site Number: 2500002, Toulouse
- Germany (2):
  - Investigational Site Number: 2760002, Minden, Northwest
  - Investigational Site Number: 2760004, Kiel
- Japan (8):
  - Investigational Site Number: 3920007, Kashiwa, Chiba
  - Investigational Site Number: 3920005, Ōita, Oita Prefecture
  - Investigational Site Number: 3920006, Hamamatsu, Shizuoka
  - Investigational Site Number: 3920004, Bunkyō City
  - Investigational Site Number: 3920003, Hamamatsu
  - Investigational Site Number: 3920009, Hirosaki
  - Investigational Site Number: 3920001, Morioka
  - Investigational Site Number: 3920002, Nishinomiya
- Poland (7):
  - Investigational Site Number: 6160002, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number: 6160001, Krakow
  - Investigational Site Number: 6160005, Lublin
  - Investigational Site Number: 6160006, Sopot
  - Investigational Site Number: 6160008, Warsaw
  - Investigational Site Number: 6160003, Warsaw
  - Investigational Site Number: 6160004, Wroclaw
- Spain (3):
  - Investigational Site Number: 7240002, Madrid
  - Investigative Site: 7240001, Madrid
  - Investigational Site Number: 7240003, Seville
- United Kingdom (5):
  - Investigational Site Number: 8260007, Bury
  - Investigational Site Number: 8260004, Cambridge
  - Investigational Site Number: 8260005, London
  - Investigational Site Number: 8260002, London
  - Investigational Site Number: 8260001, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- See also: DRI18450 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26749&tenant=MT_SNY_9011